CLINICAL TRIAL: NCT04646694
Title: The Ketamine for Acute Postoperative Analgesia (KAPA) Trial
Acronym: KAPA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-5064
Record Dates: First submitted 2020-11-17; First posted 2020-11-30 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Pain
Keywords: Postoperative; pain; effective; safe; Ketamine; placebo
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: This study will be a two arm, randomized controlled trial with a target enrollment of forty patients. Randomization will be performed with a 1:1 allocation with Ketamine or Placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The KAPA trial will be a single center, blinded (participant, caregiver, investigator, outcome assessor), parallel arm, randomized controlled feasibility trial of patients undergoing spine surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group 1 (Experimental): Patient will receive Ketamine at a dose of 30 mg every eight hours. It will be mixed with apple juice prior to administration and taken orally. Patients will receive Ketamine for three days or nine doses total.
  Interventions: Drug: Ketamine
- Study group 2 (Placebo Comparator): Patient will receive Placebo at a matching dose every eight hours. It will be mixed with apple juice prior to administration and taken orally. Patients will receive Placebo for three days or nine doses total.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ketamine — The use of oral Ketamine in this study is experimental.This study will look at how effective and safe Ketamine.
  Other Names: Ketamine Group
  Arms: Study Group 1
Other: Placebo — A placebo is given in this study to reduce the chances of believing that pain after surgery is getting better because one is receiving oral Ketamine
  Other Names: Placebo group
  Arms: Study group 2

SUMMARY:
Postoperative pain remains an important challenge for both patients and clinicians. Despite advances in pain management techniques, many patients continue to describe their pain as moderate to severe immediately after surgery. Poor postoperative pain control is associated with increased morbidity, functional impairment, and higher health care costs. While opioids currently represent the mainstay of treating surgical pain, their use is associated with significant side effects including respiratory depression, delayed recovery of bowel function as well as the potential for long-term use. Therefore, there is an urgent need to find new pain relievers with a safer side effect profiles. One such drug that has been receiving increasing attention is ketamine. Previous studies have focused on using intravenous ketamine postoperatively which requires a monitored setting but have ignored the oral form. By using the oral route of administration, ketamine could potentially be used by patients in a less resource-intensive manner with similar efficacy. Therefore, Investigators propose to conduct the Ketamine for Acute Postoperative Analgesia (KAPA) pilot study to examine the role of oral ketamine in improving recovery after spine surgery.

DETAILED DESCRIPTION:
Pain after surgery remains an important challenge for both patients and clinicians. Despite advances in pain management techniques, many patients continue to describe their pain as moderate to severe immediately after surgery. Poor surgical pain control is associated with increased morbidity, functional impairment, and higher health care costs. While opioids currently represent the mainstay of treating surgical pain, their use is associated with significant side effects including respiratory depression, delayed recovery of bowel function as well as the potential for long-term use.

Therefore, there is an urgent need to find new pain relievers with a safer side effect profiles. One such drug that has been receiving increasing attention is ketamine. Previous studies have focused on using intravenous ketamine postoperatively which requires a monitored setting but have ignored the oral form. By using the oral route of administration, ketamine could potentially be used by patients in a less resource-intensive manner with similar efficacy. Therefore, Investigators propose to conduct the Ketamine for Acute Postoperative Analgesia (KAPA) pilot study to examine the role of oral ketamine in improving recovery after spine surgery.

The drug being studied in this trial is called Ketamine. Ketamine was initially developed as a unique anesthetic drug in the 1950's, clinicians later realized that when given in low doses, Ketamine can improve pain control after surgery and other chronic neuropathic conditions. It can be particularly helpful for patients whose pain is not adequately controlled with commonly used pain medications. Ketamine has also found new roles to aid in opioid tapering of subjects with opioid dependence and in the treatment of addiction.

Health Canada has approved Ketamine for medical use in hospital setting as an IV anesthetic agent for surgical procedures. However, there are currently no Health Canada approved oral Ketamine formulations. Although, it should be noted that oral ketamine is routinely used as part of standard order sets at several health institutions across Toronto and Canada.

The use of oral Ketamine in this study is experimental. Experimental means Health Canada has not approved the oral use of Ketamine but they have approved its use in this research study.

This study will look at how effective and safe Ketamine.

If participant decide to participate, the investigator will be in contact with your regular health care provider throughout the time that you are in the study and afterwards, if needed.

Participants are being asked to take part in this research study because they will be having elective spine surgery under general anesthesia and participants may develop pain after surgery.

The usual treatment for established pain after surgery is an approved intravenous opioid, such as hydromorphone, acetaminophen and nonsteroidal anti-inflammatory drugs (NSAIDs). However, opiates usage carries significant risk of addiction and overdose, particularly with prolonged or increased dosing. Using a combination of medications to treat postoperative pain is quickly becoming more common in an attempt to avoid severe post-operative pain. Because of these limitations, it is important that Investigators look for new options to treat surgical pain.

Approximately 40 people will take part in this study at Toronto Western Hospital/UHN. Investigators expect the study to last for about 12 months.

ELIGIBILITY:
Inclusion criteria

1. Patients aged 18-75 undergoing multi-level lumbar fusion and decompression
2. Planned overnight admission to hospital

Exclusion criteria

1. Patients taking greater than 90 milligram morphine equivalents
2. History of substance use disorder
3. Previous surgery within six months
4. Pre-existing renal or liver impairment
5. Chronic benzodiazepine use
6. Psychiatric disorder with current/active pharmacologic treatment
7. Inability to complete questionnaires

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Recovery After Surgery | 30 days
  The Quality of Recovery-15 is a self-reported, patient centered outcome metric. The questionnaire has been psychometrically tested and validated. It has been shown to have good content validity, internal consistency and reliability. It captures five domains of recovery after surgery including pain, physical independence, psychological support and emotional state. It can be printed on a single sheet of paper and is easily administered in under three minutes. A change in 8 points on the score has been defined as the minimally important clinical difference in a previous study.

SECONDARY OUTCOMES:
Opioid Use | 30 days
  Opioid use as an inpatient will be determined by examining the medical administration record. During outpatient follow-up phone calls patients will be asked for their average daily opioid use. This will then be converted to a daily morphine equivalent dose.
Pain Intensity | 30 days
  Participants will use a numeric rating scale to rate their pain from 0-10. Patients will be asked to rate the maximum, minimum and average pain intensity over the past 24 hours.
Pain Interference | 30 days
  The impact of pain as measured by interference with daily activities will be measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) pain interference questionnaire.
Mood | 3 days
  Patient Health Questionaire-9 (PHQ-9) is a validated, brief diagnostic and severity measure of depression. It is sensitive to change over time and can track responses to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dinsmore, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- TWH/UHN, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No